CLINICAL TRIAL: NCT05708222
Title: Investigation of the Likelihood of a Current Major Depressive Episode in Individuals Referred to Sleep Clinics for Polysomnography (PSG) Assessment Using the MEB-001 Device.
Brief Title: Sleep Signal Analysis for Current Major Depressive Episode (SAMDE)
Acronym: SAMDE
Status: Completed | Type: Observational
Sponsor: Medibio Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-0089
Record Dates: First submitted 2022-09-25; First posted 2023-02-01 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Depressive Episode; Depression; Depressive Disorder; Depressive Disorder, Major; Depression Mild
Keywords: Major Depressive Episodes; Depression; Sleep Study
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Self Reported Assessment: This group of patients will self report their answers to the MINI assessment.
  Interventions: Device: MEB-001
- Clinician Interview Assessment: This group of patients will complete the MINI assessment via an interactive interview conducted by a qualified clinician.
  Interventions: Device: MEB-001

INTERVENTIONS:
Device: MEB-001 — The study is for the development of a software medical device. The study participant will complete study specific questionnaires and undergo a routine sleep study. The medical device will not provide any treatment or interventions.

SUMMARY:
The objective of this study is to collect data to finalize the development of MEB-001 software as a medical device. The data collected in this study will be used to develop MEB-001 machine learning algorithms by training the algorithms to match the patient's demographic and clinical information, and the objective physiological signals (i.e., electroencephalogram (EEG) and electrocardiogram (ECG)) recorded during PSG with the diagnosis of cMDE performed through the MINI neuropsychiatric evaluation.

DETAILED DESCRIPTION:
This is a two (2)-phase, single-arm, prospective, non-significant risk, multi-center trial where each enrolled subject's data will be used for the development of MEB-001.

Study Population:

Subjects who are at least 22 years old but not older than 75 years old, who have been referred to a sleep clinic for sleep disturbances and sign an informed consent form (ICF) will be evaluated for participation in this study.

The selection of the population involved in the study will consider the geographic diversity needed to obtain a representative sample of the intended use population. Centers will be selected to secure geographic and clinical diversity across the USA to obtain a representative distribution of the intended patient population.

All patients undergoing PSG due to primary or secondary sleep disorders, which include, but are not limited to, Sleep-Related Movement Disorders, Sleep-Related Breathing Disorders, Intrinsic and Extrinsic Circadian Rhythm Sleep-Wake Disorders, Hypersomnia, Parasomnia, and Insomnia, will be consecutively recruited, according to the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL the following conditions to be eligible to participate in the study:

1. Subject is age ≥ 22 years and ≤ 75 years.
2. Subject is undergoing polysomnography due to suspected primary or secondary sleep disorders.
3. Subject is willing and able to provide informed consent.
4. Subject has the ability to read and understand the instructions for the study.
5. Subject is willing to adhere to study procedures.
6. Subject is willing to undergo full night diagnostic PSG study, as prescribed.

Exclusion Criteria:

Subjects will not be eligible, and they will not be recruited to participate in the study if any of the following conditions are present:

1. Subject has a pacemaker.
2. Subject has undergone a heart transplant.
3. Subject is undergoing a full night C-PAP titration study.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are at least 22 years old but not older than 75 years old, who have been referred to a sleep clinic for sleep disturbances and sign an informed consent form (ICF) will be evaluated for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 715 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Development of software as a medical device for the assessment of current major depressive episodes. | 24 months
  Evaluation of patient objective and subjective measures to develop algorithm to determine whether the patient is experiencing a current major depressive episode.

CONTACTS AND LOCATIONS:
Overall Officials: Archie Defillo, MD, Study Chair — Medibio Limited; Melissa E Bruner, MS, Study Director — Medibio Limited
Locations (13):
- United States (13):
  - Medbridge Healthcare, Bradenton, Florida
  - Lakeland Sleep Store, Blaine, Minnesota
  - Lakeland Sleep, Plymouth, Minnesota
  - Medbridge Healthcare, Clayton, North Carolina
  - Medbridge Healthcare, Raleigh, North Carolina
  - Medbridge Healthcare, Wilson, North Carolina
  - Ohio Sleep Solutions, Columbus, Ohio
  - Ohio Sleep Solutions, Grove City, Ohio
  - Medbridge Healthcare, North Charleston, South Carolina
  - Medbridge Healthcare, Sumter, South Carolina
  - Comprehensive Sleep Medicine Associates, Austin, Texas
  - Comprehensive Sleep Medicine Associates, Sugar Land, Texas
  - Comprehensive Sleep Medicine Associates, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Caldirola D, Dacco S, Cuniberti F, Grassi M, Alciati A, Torti T, Perna G. First-onset major depression during the COVID-19 pandemic: A predictive machine learning model. J Affect Disord. 2022 Aug 1;310:75-86. doi: 10.1016/j.jad.2022.04.145. Epub 2022 Apr 27. PMID 35489559
- [Result] Caldirola D, Cuniberti F, Dacco S, Grassi M, Torti T, Perna G. Predicting New-Onset Psychiatric Disorders Throughout the COVID-19 Pandemic: A Machine Learning Approach. J Neuropsychiatry Clin Neurosci. 2022 Summer;34(3):233-246. doi: 10.1176/appi.neuropsych.21060148. Epub 2022 Mar 21. PMID 35306830
- [Result] Perna G, Dacco S, Alciati A, Cuniberti F, De Berardis D, Caldirola D. Childhood maltreatment history for guiding personalized antidepressant choice in major depressive disorder: Preliminary results from a systematic review. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Apr 20;107:110208. doi: 10.1016/j.pnpbp.2020.110208. Epub 2020 Dec 15. PMID 33338557
- [Result] Dacco S, Caldirola D, Grassi M, Alciati A, Perna G, Defillo A. High prevalence of major depression in US sleep clinics: the need for routine depression screening in sleep services. J Clin Sleep Med. 2023 Apr 1;19(4):835-836. doi: 10.5664/jcsm.10398. PMID 36644846
- [Result] Perna G, Alciati A, Dacco S, Grassi M, Caldirola D. Personalized Psychiatry and Depression: The Role of Sociodemographic and Clinical Variables. Psychiatry Investig. 2020 Mar;17(3):193-206. doi: 10.30773/pi.2019.0289. Epub 2020 Mar 12. PMID 32160691
- [Result] Perna G, Cuniberti F, Dacco S, Nobile M, Caldirola D. Impact of respiratory protective devices on respiration: Implications for panic vulnerability during the COVID-19 pandemic. J Affect Disord. 2020 Dec 1;277:772-778. doi: 10.1016/j.jad.2020.09.015. Epub 2020 Sep 7. PMID 33065816